CLINICAL TRIAL: NCT06381089
Title: The Effect of Robotic Rehabilitation and Vagus Nerve Stimulation in Addition to Robotic Rehabilitation on the Patient's Functional Level and Autonomic Nervous System in Patients With Ischemic Stroke
Brief Title: Effect Of Robotic Rehabilitation And Vagus Nerve Stimulation In Ischemia Stroke Patients
Acronym: ERRVNS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Assistant Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VNS004
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Stroke; Vagus Nerve Stimulation; Robotic Rehabilitation; Autonomic Nervous System
Keywords: Vagus Nerve Stimulation; Transcutaneous; Robotic Rehabilitation; Ischemic Stroke; Superficial EMG
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Rehabilitation Group (RRG) (Experimental): A 6-week protocol will be applied in the study. In addition to the neurological rehabilitation program, robotic rehabilitation will be applied to the RRG group 2 days a week.
  Some evaluations will be made by the researcher at two different time periods throughout the study. These time periods will be planned and carried out immediately before the study and after the 6-week treatment.
  Interventions: Device: Robotic Rehabilitation
- Vagal Nerve Stimulation With Robotic Rehabilitation Group (VRRG) (Experimental): In addition to the neurological rehabilitation program, the VRRG group will receive both robotic rehabilitation and t-VNS 2 days a week. Some evaluations will be made by the researcher at two different time periods throughout the study. These time periods will be planned and carried out immediately before the study and after the 6-week treatment.
  Interventions: Device: Robotic Rehabilitation; Device: Transcutaneous Auricular Vagal Nerve Stimulation

INTERVENTIONS:
Device: Robotic Rehabilitation — Lokomat is an exoskeleton type robotic walking device that can support both extremities symmetrically.
Device: Transcutaneous Auricular Vagal Nerve Stimulation — Vagus nerve stimulation is defined as any technique that stimulates the vagus nerve in our body.
  Arms: Vagal Nerve Stimulation With Robotic Rehabilitation Group (VRRG)

SUMMARY:
This study was conducted in patients with ischemic stroke; This study was conducted to examine the effect of robotic rehabilitation and transcutaneous auricular vagal nerve stimulation applied in addition to robotic rehabilitation on the patient's functional level and autonomic nervous system.

40 people over the age of 18 participated in the study. They were randomly divided into two groups: robotic rehabilitation and transcutaneous auricular vagal nerve stimulation applied in addition to robotic rehabilitation. While the robotic rehabilitation group received Lokomat and neurological rehabilitation, the other group received stimulation with the Vagustim device, which is applied non-invasively through the ear, in addition to Lokomat and neurological rehabilitation. Spasticity, autonomic nervous system, walking speed, motor function, quality of life, muscle activity and pain were evaluated in both groups before starting treatment and six weeks after treatment. In the study, significance was evaluated at p<0.05 level.

DETAILED DESCRIPTION:
A study group was formed, consisting of individuals who had an ischemic stroke over the age of 18, who complied with the research criteria and who signed the voluntary consent form. Age, gender, height, weight, body mass index, dominant side, affected side and time since stroke of the participants who met the inclusion criteria were recorded and randomly divided into 2 groups.

The groups are; They were divided into Robotic Rehabilitation (RRG) (n=20, 11 women, 9 men) and Transcutaneous Auricular Vagal Nerve Stimulation (VRRG) applied in addition to Robotic Rehabilitation (n=20, 9 women, 11 men) groups.

A 6-week protocol was applied in the study. In addition to the neurological rehabilitation program, robotic rehabilitation was applied to the RRG group 2 days a week. In addition to the neurological rehabilitation program, both robotic rehabilitation and transcutaneous auricular vagal nerve stimulation were applied to the VRRG group 2 days a week. Some evaluations were made by the researcher at two different time periods throughout the study. Evaluation times; T0 (before robotic rehabilitation/vagal nerve stimulation application in addition to robotic rehabilitation), T1 (robotic rehabilitation/after vagal nerve stimulation application applied in addition to robotic rehabilitation). These time periods were planned and carried out immediately before the study and after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with ischemic stroke
* Having a stroke for the first time
* Having hemiparesis
* ≤ 6 months after stroke
* Being able to walk with or without support
* Understanding and focusing on Lokomat exercises and being able to do them
* Having received walking training with Lokomat in our hospital
* Having signed the voluntary consent form
* Being over 18 years of age

Exclusion Criteria:

* Body weight more than 135 kg
* The person's height is more than two meters
* Femur length outside the range of 35-47 cm
* Intolerable leg length differences
* Peripheral nerve injury
* Peripheral neuropathy
* Anticholinergic drug use
* Presence of skin lesions
* Spasticity that prevents the locomotive from working
* Having diagnosed psychiatric problems
* Severe contracture in lower extremity muscles
* Not being able to walk before stroke
* Having a history of additional neurological diseases (Parkinson, etc.)
* Unstable cardio-pulmonary disease
* Having orthopedic fractures (lower extremity fractures) and/or joint implants
* Severe osteoporosis
* Uncontrolled hypertension despite medication use
* Lower extremity amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | Time Frame: within 10 minutes after intervention
  Numerical pain scale is used to classify pain from 0 to 10. '0' means no pain and '10' means unbearable pain.
Stroke Specific Quality of Life Scale | Time Frame: within 10 minutes after intervention
  The stroke-specific quality of life scale consists of a total of 49 items in 12 domains. Each item is scored between 1 (strongly agree) and 5 (strongly disagree). The total score is evaluated between 49 and 245 points. A score of 49 indicates the lowest quality of life and 245 indicates the highest quality of life.
10 Meter Walk Test | Time Frame: within 10 minutes after intervention
  During the test, the patient's walking performance is recorded in terms of time between two markers located 10 meters apart. It is used to determine functional mobility and walking speed.
Fugl-Meyer Assessment Lower Extremity | Time Frame: within 10 minutes after intervention
  It is a widely used scale in the evaluation of motor function after stroke. The lower extremity section consists of 17 items and its maximum score is 34 points.
Modified Ashworth Scale | Time Frame: within 10 minutes after intervention
  It is the universally accepted clinical tool used to measure increases in muscle tone.
Electromyography | Time Frame: within 10 minutes after intervention
  It refers to the collective electrical signals during the contraction of muscles connected to the nervous system. EMG devices evaluate and interpret the electrical potential that enables the contraction of voluntary muscles. The EMG device evaluates voluntarily working skeletal muscles. EMG, a muscle examination, monitors and interprets the electrical activity that causes muscles to contract. EMG examinations are defined as a set of tests that include nerve examination as well as examination of muscle activation.
Autonomic Nervous System | Time Frame: within 10 minutes after intervention
  The Polar H10 device is a gold-standard HRV sensor of high sensitivity and accuracy that comes with a wearable chest strap. The device comes with a soft, adjustable sensor that contacts the chest to capture HRV in real time.

CONTACTS AND LOCATIONS:
Overall Officials: SEFA HAKTAN HATIK, PhD, Study Chair — Sinop University